CLINICAL TRIAL: NCT04865627
Title: Accuracy of Activity Monitors Based on Accelerometers and/or Multiple Sensors for the Objective Measurement of Physical Activity of Geriatric Patients During Hospitalization in Acute Care of Elderly (ACE) and Geriatric Rehabilitation Units
Brief Title: Accuracy Activity Monitors for Inhospital Activity Monitoring of Geriatric Patients
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Margaretha van Dijk, Physiotherapist, KU Leuven
Other Study IDs: S64932
Record Dates: First submitted 2021-04-21; First posted 2021-04-29 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Hip Fractures; Stroke; Abdominal Injury
Keywords: geriatric inhospital rehabilitation; elderly; activity monitors
MeSH Terms: conditions — Hip Fractures; Stroke; Abdominal Injuries | interventions — Fitness Trackers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- independent walking with walking aid: the participant is able to walk with a walking aid and does not need further assistance.
  Interventions: Device: activity monitor
- dependent walking with walking aid: the participant is able to walk with assistance and a walking aid
  Interventions: Device: activity monitor

INTERVENTIONS:
Device: activity monitor — Both groups will wear three different activity monitors for one week. There is one observation moment which consists of four minutes lying, sitting, standing, walking and taking stairs. Participants will be filmed during this moment.
  Other Names: accelerometer; activity sensor

SUMMARY:
The focus of this study will be to determine the accuracy of the MOX, the Axivity and Fitbit, Empatica and Chill+ activity monitors (with both custom-made and available algorithms) for the classification of lying, sitting, standing, walking and climbing stairs in hospitalized older people in Acute Care for the elderly (ACE) and geriatric rehabilitation units.

In addition, the feasibility of the use of the activity monitors as a measurement tool in daily practice during hospitalization in the geriatric department will be investigated.

DETAILED DESCRIPTION:
Adequate physical activity and exercise throughout the day are important to maximize independence and quality of life. To be able to optimize the physiotherapeutic interventions and to monitor how much geriatric patients move during hospitalization, it is desirable to follow up their activity by means of an activity monitor. In this study the investigators will determine the accuracy of three different types of activity monitors, the "MOX" placed on the thigh, the "Axivity" placed on the torso and the "Fitbit Sense", the "Empatica" and the "Chill+" placed on the wrist, for the classification of lying, sitting, standing, walking and climbing stairs in hospitalized older people in the geriatric department.

In this clinical study, 40 patients will participate of which 20 hospitalized in the geriatric rehabilitation unit at campus Pellenberg and 20 hospitalized in the acute care of elderly units at campus Gasthuisberg UZ Leuven, Belgium.

These activity monitors will remain attached for seven days so that activity can monitored during the week as well as on weekends. In an experimental test session a total of five activities (lying down, sitting, standing, walking and possibly climbing stairs) will be performed and observed, each lasting four minutes. The observations will be recorded by video where only the lower body will be in focus.

There will be daily checks to see if the activity monitors on the thigh, torso, and wrist stay in place, if the skin tolerates it well, if participants experiencing subjective discomfort, and if the measurements continue. At the end of the week, a short questionnaire will be completed on the user-friendliness of the different monitors.

The investigators will use the accuracy and patient satisfaction outcomes to decide the feasibility of using these activity monitors as a measurement tool in daily practice during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the rehabilitation or acute ward of UZ Leuven
* walking with the use of a walkingaid
* a signed informed consent form
* an expected stay of at least 7 days

Exclusion Criteria:

* medically unstable

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Participant are admitted to a geriatric ward in UZ Leuven, Belgium and use a walkingaid.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
accuracy of the activity monitors compared to the observation | 30 minutes
  accuracy of the activity monitors during the observation moment, second by second

SECONDARY OUTCOMES:
usability of an activity monitor in daily practice on the ward | one week
  Short questionnaire to explore the usability of the activity monitors

CONTACTS AND LOCATIONS:
Overall Officials: Johan Flamaing, MD, PhD, Principal Investigator — UZ Leuven, KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium

REFERENCES:
- [Result] van Dijk M, Bijnens W, Van Driessche C, Van Meerbeek T, Allegaert P, Van Cleynenbreugel H, Verschueren S, Verheyden G, Tournoy J, Flamaing J. Accuracy of an Activity Monitor in Assessing Physical Activity of Hospitalized Geriatric Rehabilitation Patients With Slow Walking Speed Using a Walking Aid. J Aging Phys Act. 2024 Nov 20;33(3):243-250. doi: 10.1123/japa.2023-0319. Print 2025 Jun 1. PMID 39566489